CLINICAL TRIAL: NCT03231059
Title: GLOBAL LEADERS Adjudication Sub-Study
Acronym: GLASSY
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: European Cardiovascular Research Center (Network)
Responsible Party: Sponsor
Other Study IDs: 039_2013_Substudy
Record Dates: First submitted 2017-07-19; First posted 2017-07-27 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Coronary Artery Disease; Platelet-aggregation Inhibitors
Keywords: Coronary artery disease; Percutaneous coronary intervention; Drug-eluting stent; Antiplatelet drugs; Clinical event committee
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental treatment strategy: All patients in the treatment group received acetylsalicylic acid (ASA) and ticagrelor for 1 month followed by 23 months of ticagrelor monotherapy
- Reference treatment strategy: Acute Coronary Syndrome (ACS) patients incl. unstable angina (UA) patients: ASA and ticagrelor for 12 months followed by 12 months of ASA monotherapy.
  Stable Coronary Artery Disease (CAD) patients: ASA and clopidogrel for 12 months followed by 12 months of ASA monotherapy.

SUMMARY:
The GLOBAL LEADERS Adjudication Sub-StudY, GLASSY, is based on a re-assessment of all the events reported in the dataset of the parent trial (COMPARATIVE EFFECTIVENESS OF 1 MONTH OF TICAGRELOR PLUS ASPIRIN FOLLOWED BY TICAGRELOR MONOTHERAPY VERSUS A CURRENT-DAY INTENSIVE DUAL ANTIPLATELET THERAPY IN ALL-COMERS PATIENTS UNDERGOING PERCUTANEOUS CORONARY INTERVENTION WITH BIVALIRUDIN AND BIOMATRIX FAMILY DRUG-ELUTING STENT USE) by an independent Clinical Event Committee (CEC), composed of three physicians not involved in the main trial. The substudy include the first 19 top-enrolling sites of the GLOBAL LEADERS to reach the estimated sample size of 7,186 patients for the two co-primary outcomes of death, any non-fatal myocardial infarction, any non-fatal stroke or urgent target vessel revascularization and bleeding events classified as 3 or 5 according to the Bleeding Academic Research Consortium (BARC) criteria. To ensure a comprehensive assessment of clinical events, a triggers logic is adopted to identify other potential events qualifying for study endpoints but not reported as such by local investigators.

DETAILED DESCRIPTION:
The GLOBAL LEADERS trial was designed to determine the benefits and risks of an antithrombotic regimen using ticagrelor 90 mg BID combined with low-dose (75 mg OD) acetylsalicylic acid (ASA) for one month followed by ticagrelor 90 mg BID alone for 23 months, compared to conventional dual antiplatelet therapy (DAPT) in all-comers patients with coronary artery disease undergoing biolimus-eluting stent implantation on bivalirudin. It was intended as a pragmatic clinical trial and, by design, endpoints included in primary and secondary analyses are only investigator-reported (IR) and will not undergo independent adjudication by a CEC. It is well known that in the absence of blinding of randomized treatment (i.e. in an open-label design such as GLOBAL LEADERS) the use of IR outcome may introduce detection and/or reporting bias. There are multiple lines of evidence indicating that central and independent adjudication of events may affect the results of a randomized trial by minimizing variability and heterogeneity inherently present when several different clinicians and data managers apply definitions of endpoints which are complex and sometimes not well known.Moreover, independent adjudication of ischaemic and bleeding endpoints may provide important mechanistic information that may deepen understanding of the primary endpoint result of the study by better characterizing component of such endpoints including, but not limited to, precise cause of death, sub-type of myocardial infarction (MI), and bleeding location. The objectives of this substudy are: to assess the impact of CEC-adjudication process on the results of the study; to quantify the added value of CEC adjudication process for endpoint reporting by evaluating the concordance between IR-reported and CEC-adjudicated events; to gather mechanistic information to aid in the interpretation of the effect of the experimental treatment in the parent trial and to identify specific subgroups of patients that could particularly benefit from the experimental therapy in terms of ischemic and bleeding events.

ELIGIBILITY:
Inclusion Criteria:

"All comer" patients

1. Age ≥18 years;
2. Presence of one or more coronary artery stenoses of 50% or more in a native coronary artery or in a saphenous venous or arterial bypass conduit suitable for coronary stent implantation. The vessel should have a reference vessel diameter of at least 2.25 mm (no limitation on the number of treated lesions, vessels, or lesion length);
3. Able to provide informed consent and willing to participate in 2 year follow- up period.

Exclusion Criteria:

1. Known intolerance to aspirin, P2Y12 inhibitors, bivalirudin, stainless steel or biolimus;
2. Known intake of a strong CYP3A4 inhibitor (e.g., ketoconazole, clarithromycin, nefazodone, ritonavir, and atazanavir), as co-administration may lead to a substantial increase in exposure to ticagrelor;
3. Known moderate to severe hepatic impairment (alanine-aminotransferase ≥ 3 x ULN);
4. Planned surgery, including CABG as a staged procedure (hybrid) within 12 months of the index procedure, unless dual antiplatelet therapy is maintained throughout the peri-surgical period;
5. Need for chronic oral anti-coagulation therapy;
6. Active major bleeding or major surgery within the last 30 days;
7. Known history of intracranial haemorrhagic stroke or intra-cranial aneurysm;
8. Known stroke (any type) within the last 30 days;
9. Known pregnancy at time of randomisation;
10. Female who is breastfeeding at time of randomisation;
11. Currently participating in another trial and not yet at its primary endpoint

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients included in the GLOBAL LEADERS Trial, e.g. "All comers" with coronary artery disease requiring percutaneous coronary intervention (PCI)
Sampling Method: Non-Probability Sample
Enrollment: 7365 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Composite of death, stroke, cardiac and bleeding events | 24 months
  Death, any non-fatal MI, any non-fatal stroke (i.e. including both ischemic and haemorrhagic) or urgent target vessel revascularization (TVR) (co-primary efficacy endpoint) Bleeding 3 or 5 according to Bleeding Academic Research Consortium (BARC) definition (co-primary safety endpoint).
  Primary outcome will be defined as the occurrence of the sum of listed events

SECONDARY OUTCOMES:
Death | 24 months or at earlier time point
  Any death
Non-fatal MI | 24 months or at earlier time point
  Any non-fatal MI
Non-fatal stroke | 24 months or at earlier time point
  Any non-fatal stroke (i.e. including both ischemic and haemorrhagic)
Rates of urgent revascularization of the target vessel (Urgent TVR) | 24 months or at earlier time point
  One or more episodes of rest pain, presumed to be ischemic in origin which results in either urgent percutaneous coronary intervention or urgent coronary artery by pass graft. To be considered urgent, the repeat revascularization will be initiated within 24 hours of the last episode of ischemia and not be identified as planned or staged.
Definite, probable or possible Stent thrombosis | 24 months or at earlier time point
  Definite, probable or possible Stent thrombosis according to Academic Research Consortium (ARC) classification
Bleeding events | 24 months or at earlier time point
  Bleeding events according to Bleeding Academic Research Consortium (BARC), Thrombolysis In Myocardial Infarction (TIMI) and Global Use of Strategies To Open coronary arteries (GUSTO) classifications
Differences between the rates of outcomes reported by the investigators and the rates of outcomes as adjudicated by an independent clinical event committee | 24 months or at earlier time point
  Concordance between IR- and CEC- endpoints

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Windecker, MD, Study Chair — Inselspital Bern University Hospital; Marco Valgimigli, MD, Principal Investigator — Inselspital Bern University Hospital
Locations (19):
- Wilhelminenspital 1160, Vienna, Austria
- Belgium (4):
  - Research centre Bonheiden 3204, Bonheiden
  - Research centre Charleroi 3202, Charleroi
  - Research centre Genk 3205, Genk
  - Research centre Hasselt 3203, Hasselt
- Research centre Sofia, 9901, Sofia, Bulgaria
- Germany (2):
  - Research centre Bad Nauheim 4902, Bad Nauheim
  - Research centre Essen 4903, Essen
- Italy (4):
  - Research centre Arezzo 3902, Arezzo
  - Research centre Ferrara 3905, Ferrara
  - Research centre Pavia 3903, Pavia
  - Research centre Terni 3909, Terni
- Netherlands (2):
  - Research centre Amsterdam 3104, Amsterdam
  - Research centre Rotterdam 3101, Rotterdam
- Poland (3):
  - Research centre Chrzanow 4802, Chrzanów
  - Research centre Dabrowa Gornicza 4801, Dąbrowa Górnicza
  - Research centre Krakov 4807, Krakow
- Inselspital Bern University Hospital, Bern, Switzerland
- Research centre Blackburn 4404, Blackburn, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vranckx P, Valgimigli M, Windecker S, Steg PG, Hamm C, Juni P, Garcia-Garcia HM, van Es GA, Serruys PW. Long-term ticagrelor monotherapy versus standard dual antiplatelet therapy followed by aspirin monotherapy in patients undergoing biolimus-eluting stent implantation: rationale and design of the GLOBAL LEADERS trial. EuroIntervention. 2016 Nov 20;12(10):1239-1245. doi: 10.4244/EIJY15M11_07. PMID 26606735
- [Background] Seltzer JH, Turner JR, Geiger MJ, Rosano G, Mahaffey KW, White WB, Sabol MB, Stockbridge N, Sager PT. Centralized adjudication of cardiovascular end points in cardiovascular and noncardiovascular pharmacologic trials: a report from the Cardiac Safety Research Consortium. Am Heart J. 2015 Feb;169(2):197-204. doi: 10.1016/j.ahj.2014.11.003. Epub 2014 Nov 10. PMID 25641528
- [Background] Lopes RD, Dickerson S, Hafley G, Burns S, Tourt-Uhlig S, White J, Newby LK, Komajda M, McMurray J, Bigelow R, Home PD, Mahaffey KW. Methodology of a reevaluation of cardiovascular outcomes in the RECORD trial: study design and conduct. Am Heart J. 2013 Aug;166(2):208-216.e28. doi: 10.1016/j.ahj.2013.05.005. Epub 2013 Jun 22. PMID 23895802
- [Background] Vranckx P, McFadden E, Cutlip DE, Mehran R, Swart M, Kint PP, Zijlstra F, Silber S, Windecker S, Serruys PW. Clinical endpoint adjudication in a contemporary all-comers coronary stent investigation: methodology and external validation. Contemp Clin Trials. 2013 Jan;34(1):53-9. doi: 10.1016/j.cct.2012.08.012. Epub 2012 Sep 10. PMID 22975439
- [Background] Vranckx P, McFadden E, Mehran R, Cutlip DE. Clinical event committees in coronary stent trials: insights and recommendations based on experience in an unselected study population. EuroIntervention. 2012 Jul 20;8(3):368-74. doi: 10.4244/EIJV8I3A56. PMID 22829511
- [Background] Mahaffey KW, Wampole JL, Stebbins A, Berdan LG, McAfee D, Rorick TL, French JK, Kleiman NS, O'Connor CM, Cohen EA, Granger CB, Armstrong PW; APEX-AMI Investigators. Strategic lessons from the clinical event classification process for the Assessment of Pexelizumab in Acute Myocardial Infarction (APEX-AMI) trial. Contemp Clin Trials. 2011 Mar;32(2):178-87. doi: 10.1016/j.cct.2010.12.013. Epub 2011 Jan 8. PMID 21220052
- [Background] Frederich R, Alexander JH, Fiedorek FT, Donovan M, Berglind N, Harris S, Chen R, Wolf R, Mahaffey KW. A systematic assessment of cardiovascular outcomes in the saxagliptin drug development program for type 2 diabetes. Postgrad Med. 2010 May;122(3):16-27. doi: 10.3810/pgm.2010.05.2138. PMID 20463410
- [Background] Kirwan BA, Lubsen J, de Brouwer S, Danchin N, Battler A, Bayes de Luna A, Dunselman PH, Glasser S, Koudstaal PJ, Sutton G, van Dalen FJ, Poole-Wilson PA; ACTION (A Coronary disease Trial Investigating Outcome with Nifedipine GITS) investigators. Diagnostic criteria and adjudication process both determine published event-rates: the ACTION trial experience. Contemp Clin Trials. 2007 Nov;28(6):720-9. doi: 10.1016/j.cct.2007.04.001. Epub 2007 Apr 19. PMID 17509947
- [Background] Petersen JL, Haque G, Hellkamp AS, Flaker GC, Mark Estes NA 3rd, Marchlinski FE, McAnulty JH, Greenspon AJ, Marinchak RA, Lee KL, Lamas GA, Mahaffey KW; MOST Clinical Events Committee. Comparing classifications of death in the Mode Selection Trial: agreement and disagreement among site investigators and a clinical events committee. Contemp Clin Trials. 2006 Jun;27(3):260-8. doi: 10.1016/j.cct.2006.02.002. Epub 2006 Mar 29. PMID 16574497
- [Background] Mahaffey KW, Roe MT, Dyke CK, Newby LK, Kleiman NS, Connolly P, Berdan LG, Sparapani R, Lee KL, Armstrong PW, Topol EJ, Califf RM, Harrington RA. Misreporting of myocardial infarction end points: results of adjudication by a central clinical events committee in the PARAGON-B trial. Second Platelet IIb/IIIa Antagonist for the Reduction of Acute Coronary Syndrome Events in a Global Organization Network Trial. Am Heart J. 2002 Feb;143(2):242-8. doi: 10.1067/mhj.2002.120145. PMID 11835026
- [Background] Mahaffey KW, Harrington RA, Akkerhuis M, Kleiman NS, Berdan LG, Crenshaw BS, Tardiff BE, Granger CB, DeJong I, Bhapkar M, Widimsky P, Corbalon R, Lee KL, Deckers JW, Simoons ML, Topol EJ, Califf RM; For the PURSUIT Investigators. Disagreements between central clinical events committee and site investigator assessments of myocardial infarction endpoints in an international clinical trial: review of the PURSUIT study. Curr Control Trials Cardiovasc Med. 2001 Jul 17;2(4):187-194. doi: 10.1186/cvm-2-4-187. PMID 11806794
- [Derived] Leonardi S, Branca M, Franzone A, McFadden E, Piccolo R, Juni P, Vranckx P, Steg PG, Serruys PW, Benit E, Liebetrau C, Janssens L, Ferrario M, Zurakowski A, Diletti R, Dominici M, Huber K, Slagboom T, Buszman P, Bolognese L, Tumscitz C, Bryniarski K, Aminian A, Vrolix M, Petrov I, Garg S, Naber C, Prokopczuk J, Hamm C, Heg D, Windecker S, Valgimigli M. Comparison of Investigator-Reported and Clinical Event Committee-Adjudicated Outcome Events in GLASSY. Circ Cardiovasc Qual Outcomes. 2021 Feb;14(2):e006581. doi: 10.1161/CIRCOUTCOMES.120.006581. Epub 2021 Feb 4. PMID 33535773
- [Derived] Franzone A, McFadden EP, Leonardi S, Piccolo R, Vranckx P, Serruys PW, Hamm C, Steg PG, Heg D, Branca M, Juni P, Windecker S, Valgimigli M; Collaborators. Ticagrelor alone or conventional dual antiplatelet therapy in patients with stable or acute coronary syndromes. EuroIntervention. 2020 Oct 23;16(8):627-633. doi: 10.4244/EIJ-D-20-00145. PMID 32482616
- [Derived] Franzone A, McFadden E, Leonardi S, Piccolo R, Vranckx P, Serruys PW, Benit E, Liebetrau C, Janssens L, Ferrario M, Zurakowski A, Diletti R, Dominici M, Huber K, Slagboom T, Buszman P, Bolognese L, Tumscitz C, Bryniarski K, Aminian A, Vrolix M, Petrov I, Garg S, Naber C, Prokopczuk J, Hamm C, Steg PG, Heg D, Juni P, Windecker S, Valgimigli M; GLASSY Investigators. Ticagrelor Alone Versus Dual Antiplatelet Therapy From 1 Month After Drug-Eluting Coronary Stenting. J Am Coll Cardiol. 2019 Nov 5;74(18):2223-2234. doi: 10.1016/j.jacc.2019.08.1038. PMID 31672177